CLINICAL TRIAL: NCT07093060
Title: The Influence and Regulatory Role of Exogenous and Endogenous Oxytocin on Social Attention in Humans
Brief Title: The Effect of Oral Oxytocin and Atosiban on Social Attention
Acronym: OTAtosiban
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 106142023111727716
Record Dates: First submitted 2025-07-09; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healhty
Keywords: Oxytocin; Atosiban; Eye tracking; Autistic trait
MeSH Terms: interventions — Oxytocin; atosiban

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design experiment including 5 treatment groups receiving oral oxytocin, atosiban, or placebo interventions prior to performing visual attention tasks
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- oxytocin 24IU group (Experimental): Interventions are placebo followed after 15 min by the lower dose (24IU) oxytocin
  Interventions: Drug: Oxytocin lower dose (24IU); Drug: Placebo
- atosiban group (Experimental): Interventions are placebo followed after 15 minutes by 150ug atosiban
  Interventions: Drug: Atosiban; Drug: Placebo
- placebo group (Placebo Comparator): Interventions are placebo followed after 15 minutes by another placebo
  Interventions: Drug: Placebo
- oxytocin 48IU group (Experimental): Interventions are placebo followed after 15 minutes by the higher 48IU oxytocin dose
  Interventions: Drug: Oxytocin higher dose (48IU); Drug: Placebo
- Atosiban and 24IU oxytocin group (Experimental): Interventions are atosiban 150ug followed after 15 minutes by the lower (24IU) dose of oxytocin
  Interventions: Drug: Oxytocin lower dose (24IU); Drug: Atosiban

INTERVENTIONS:
Drug: Oxytocin lower dose (24IU) — Oxytocin (24IU) will be administered as a lingual spray (6, 0.1 puffs (4IU per puff) of spray on and under the tongue)
  Other Names: oral oxytocin 24IU
  Arms: Atosiban and 24IU oxytocin group; oxytocin 24IU group
Drug: Oxytocin higher dose (48IU) — 48IU oxytocin administered as a lingual spray (6, 0.1ml sprays (8IU per puff) on or under the tongue)
  Other Names: oral oxytocin 48IU
  Arms: oxytocin 48IU group
Drug: Atosiban — 150ug atosiban administered by lingual sprays (6, 0.1ml sprays on and under the tongue)
  Other Names: oral atosiban
  Arms: Atosiban and 24IU oxytocin group; atosiban group
Drug: Placebo — Placebo administered as a lingual spray (6, 0.1 ml sprays one and under the tongue. Placebo has the same composition of 0.9% saline and glycerol as for oxytocin and atosiban interventions
  Arms: atosiban group; oxytocin 24IU group; oxytocin 48IU group; placebo group

SUMMARY:
The main aim of the present study is to investigate whether orally (lingual spray) administered oxytocin influences human social attention and behaviors via oxytocin receptors and whether its effects are dose- and task-dependent.

DETAILED DESCRIPTION:
In a placebo-controlled double-blind between-subject design experiment, investigators plan to investigate whether oral (lingual spray) oxytocin influences human social attention and behaviors via the oxytocin receptor and whether its effects are dose- and task-dependent. Participants complete questionnaires in Chinese versions before treatment administration, including Trait Anxiety Inventory, State Anxiety Inventory, Liebowitz Social Anxiety Scale, Beck Depression Inventory, Autism Spectrum Quotient. Then the first blood (6 ml via indwelling medial cubital vein catheter) and saliva (1-2 ml, passive drool) samples are collected, followed by the first self-administered medication (three sublingual and three supragingival administrations, alternating separated by 30 seconds). After a 15-minute interval, the second medication is administered, with a second blood sample collected immediately afterwards. Participants then remain in the lab for 30 minutes (mobile phone use and conversation with experimenters prohibited during this period). Behavioral experiments commence after the third blood collection. Behavioral experiment consists of four visual attention paradigms including a dynamic task simultaneously contrasting social stimuli (individuals dancing) with geometric patterns; social directed attention using a gaze following paradigm; face emotion processing, and empathy for individuals depicted in natural scenes exhibiting strong positive or negative emotions. During these phases, participants' fixation time, fixation counts and pupil size on specified areas of interest during each visual attention paradigm will be measured using eye tracking equipment. Immediately after completion of the paradigm, participants will complete the state anxiety questionnaire again to assess treatment/paradigm effects on anxiety.

MANOVA tests followed by appropriate post-hoc analyses will be performed on eye-tracking and other data to assess treatment effects. Correlation analysis will be used to assess associations between trait autism scores and outcome measures in the different groups.

Investigators hypothesize that oral oxytocin treatment will dose-dependently facilitate enhanced interest in social stimuli or features in the different visual attention paradigms and dose-dependently increase oxytocin concentrations. Investigators additionally hypothesize that the oxytocin receptor antagonist, atosiban, will reduce interest in social stimuli or features and will prevent facilitatory effects of oxytocin administration but not influence oxytocin concentrations. Investigators hypothesize that oxytocin treatment will increase pupil diameter while viewing some of the social stimuli. Investigators hypothesize that there will be no treatment-dependent effects on state anxiety. Investigators hypothesize that oxytocin effects on enhancing social attention will be greater in individuals with higher scores on trait autism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* History of or current neurological/psychiatric disorders;
* Use of psychotropic medications (including nicotine)
* Visual impairments

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects without past or current psychiatric or neurological disorders
Enrollment: 250 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Fixation duration | Fixation durations will be taken for each of the areas of interest in the four different visual paradigms starting 45 minutes post-treatment from the beginning of each paradigm until the end of each paradigm (each paradigm lasts around 10 minutes)
  Fixation time on different areas of interest in the different visual presentation paradigms using eye-tracking
Fixation counts | Fixation counts will be taken for each of the areas of interest in the four different visual paradigms starting 45 minutes post-treatment, from the beginning of each paradigm until the end of each paradigm (each paradigm lasts around 10 minutes).
  Total number of fixations made by participant towards the different areas of interest in the different visual paradigms using eye-tracking

SECONDARY OUTCOMES:
Oxytocin concentration | Blood samples taken at time 0 (baseline), 15 minutes after first treatment, and 30 minutes after second treatment. Saliva samples taken at time 0 (baseline) and after visual paradigms (around 90 minutes post treatment).
  OT concentrations will be measured in blood (plasma) samples (6ml) taken from indwelling catheter in median cubital vein and saliva samples (1-2 ml) taken using passive drool. Oxytocin concentrations will be measured using appropriate assays.
Pupil size | Pupil size will be measured starting 45 min post-treatment during the whole of each of the different visual presentation paradigms (around 10 minutes for each paradigm).
  Pupil size will be measured while subjects view different areas of interest in different visual presentation paradigms using an eye-tracker
State anxiety | Subjects will complete the questionnaire twice, once immediately prior to treatment (baseline) and a second time immediately after completion of the four visual paradigms (around 90 minutes post treatment).
  State anxiety will be measured using a questionnaire (40 self-report question - State-Trait Anxiety Inventory, with total scores ranging from 20 to 80, where higher scores indicate greater anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared with other qualified researchers upon request